CLINICAL TRIAL: NCT02013310
Title: A Phase 2, Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing HT-0712 With Placebo in Subjects With Age-Associated Memory Impairment (AAMI)
Brief Title: HT-0712 vs. Placebo in Subjects With Age-Associated Memory Impairment (AAMI)
Acronym: PRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-0712-201
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Age-Associated Memory Impairment (AAMI)
MeSH Terms: interventions — HT-0712

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HT-0712 (50mg) (Experimental): HT-0712 capsules administered once daily.
  Interventions: Drug: HT-0712
- Placebo (Placebo Comparator): Placebo capsules administered once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HT-0712
  Arms: HT-0712 (50mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, multicenter, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy of HT-0712 in improving memory and cognitive performance in subjects with Age-Associated Memory Impairment (AAMI)

ELIGIBILITY:
Main Inclusion Criteria:

* Complaints of memory loss in everyday life
* Performance at least one standard deviation below the mean established for young adults on standardized memory tests
* Absence of dementia
* Intact global intellectual function

Main Exclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (MCI) or Alzheimer's Disease
* Evidence of dementia
* Evidence of psychiatric or neurological disorder that could influence cognition or contributed to the subject's memory loss
* Use of any drugs that could influence cognition

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Drug Research™ (CDR) Study Specific Test Battery | Weekly over the course of 6-weeks

SECONDARY OUTCOMES:
Paired Associated Learning and Memory Test | Weekly over the course of 6-weeks
Subject Global Impression Scale of Cognition (SGI-Cog) | Weekly over the course of 6-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Perera, MD, Study Director — Dart NeuroScience, LLC
Locations (16):
- United States (16):
  - Sun City, Arizona
  - Long Beach, California
  - Santa Monica, California
  - Denver, Colorado
  - Atlantis, Florida
  - Brooksville, Florida
  - Tampa, Florida
  - Marlton, New Jersey
  - Princeton, New Jersey
  - New York, New York
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Cordova, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah